CLINICAL TRIAL: NCT03797963
Title: Split-mouth Randomized Clinical Study on the Use of Symbios Xenograft for Sinus Floor Elevation
Brief Title: Clinical Study on the Use of Symbios Xenograft for Sinus Floor Elevation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Pablo Galindo-Moreno, Full Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 480CEIH2018
Record Dates: First submitted 2019-01-06; First posted 2019-01-09 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Sinus Floor Augmentation
Keywords: Maxillary sinus augmentation; Sinus lift; Biomaterial; Anorganic bovine bone; Porcine bone mineral; Implant dentistry

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBM+ACB (Active Comparator): Porcine bone mineral (Symbios Xenograft) + autogenous cortical bone
  Interventions: Device: PBM+ACB
- ABB+ACB (Experimental): Anorganic bovine bone (BioOss Xenograft) + autogenous cortical bone
  Interventions: Device: ABB+ACB

INTERVENTIONS:
Device: PBM+ACB — Maxillary sinus floor elevation and bone grafting with the use of porcine bone mineral biomaterial (Symbios Xenograft) combined with autogenous cortical bone
  Arms: PBM+ACB
Device: ABB+ACB — Maxillary sinus floor elevation and bone grafting with the use of anorganic bovine bone biomaterial (BioOss Xenograft) combined with autogenous cortical bone
  Arms: ABB+ACB

SUMMARY:
The study aims to evaluate the clinical and radiological behavior, the histological and morphometrical components, the expression of proteins related to bone formation, and the analysis of markers of reparative mesenchymal stromal cells, after using two different xenogenic biomaterials in combination with autogenous cortical bone for maxillary sinus floor elevation.

A randomized split-mouth clinical study is designed to include patients in need of two-stage bilateral maxillary sinus floor elevation. Patients will be assigned to receive a mix of autogenous cortical bone (collected by a bone scraper from the access window to the maxillary sinus) and anorganic bovine bone (BioOss Xenograft) in one maxillary sinus or autogenous cortical bone and porcine bone mineral (Symbios Xenograft) in the other maxillary sinus. Cone-beam computerized tomography (CBCT) scans will be performed before and after sinus floor elevation and 6, 12 and 18 months after the procedure to assess the bone gain. Bone core biopsies will be obtained at the site of implant placement 6 months after the floor elevation. Histological sections will be subjected to histomorphometric and immunohistochemical evaluation of differentiation markers.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous patients.
* Kennedy class I in the upper jaw.
* Less than 5 mm of residual crestal bone to the maxillary sinus.
* Need for the replacement of teeth with dental implants.

Exclusion Criteria:

* Sinus pathology (sinusitis, mucocele, cysts).
* Smokers.
* Previous long-term (>3 months) use of drugs known to affect bone metabolism, such as bisphosphonates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
Sinus floor height change | From surgery to 6 months
  CBCT scans will be performed after the sinus floor elevation and 6 months later before implant placement to calculate vertical bone height change

SECONDARY OUTCOMES:
Sinus floor height change after 12 months | From surgery to 12 months
  CBCT scans will be performed after the sinus floor elevation and 12 months later to calculate vertical bone height change
Sinus floor height change after 18 months | From surgery to 18 months
  CBCT scans will be performed after the sinus floor elevation and 18 months later to calculate vertical bone height change
Area of new mineralized tissue | 6 months
  Histomorphometric quantification of new mineralized tissue in a bone biopsy collected 6 months after the grafting procedure
Area of non-mineralized tissue | 6 months
  Histomorphometric quantification of non-mineralized tissue in a bone biopsy collected 6 months after the grafting procedure
Area of remaining graft particles | 6 months
  Histomorphometric quantification of remaining graft particles in a bone biopsy collected 6 months after the grafting procedure

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Galindo-Moreno, DDS, MS, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Universidad de Granada, Granada, Spain

REFERENCES:
- [Background] Galindo-Moreno P, de Buitrago JG, Padial-Molina M, Fernandez-Barbero JE, Ata-Ali J, O Valle F. Histopathological comparison of healing after maxillary sinus augmentation using xenograft mixed with autogenous bone versus allograft mixed with autogenous bone. Clin Oral Implants Res. 2018 Feb;29(2):192-201. doi: 10.1111/clr.13098. Epub 2017 Oct 26. PMID 29071736
- [Background] Galindo-Moreno P, Avila G, Fernandez-Barbero JE, Aguilar M, Sanchez-Fernandez E, Cutando A, Wang HL. Evaluation of sinus floor elevation using a composite bone graft mixture. Clin Oral Implants Res. 2007 Jun;18(3):376-82. doi: 10.1111/j.1600-0501.2007.01337.x. Epub 2007 Mar 12. PMID 17355356
- [Result] Galindo-Moreno P, Abril-Garcia D, Carrillo-Galvez AB, Zurita F, Martin-Morales N, O'Valle F, Padial-Molina M. Maxillary sinus floor augmentation comparing bovine versus porcine bone xenografts mixed with autogenous bone graft. A split-mouth randomized controlled trial. Clin Oral Implants Res. 2022 May;33(5):524-536. doi: 10.1111/clr.13912. Epub 2022 Mar 3. PMID 35224778